CLINICAL TRIAL: NCT00461448
Title: Pilot Study of Potassium Supplementation in the Treatment of Rheumatoid Arthritis: a 4-Week, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: A Pilot Study of Potassium Supplementation for Adult Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Reza Rastmanesh, SBMU
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NNFTRI-B2484
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Potassium supplement; Rheumatoid Arthritis; Pain; Disease Activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Potassium supplement (Active Comparator): Patients received an Enriched Grape Juice containing 234.5 mmol microcrystalline KCl (a total of 6000 mg of K in 2 EGJ, but split into 2 intakes daily)
  Interventions: Dietary Supplement: Potassium supplement
- 2 Grape Juice (Placebo Comparator): Patients received same amount of grape juice for 28 days.
  Interventions: Dietary Supplement: Potassium supplement

INTERVENTIONS:
Dietary Supplement: Potassium supplement — Patients were randomly allocated to receive either an EGJ containing 234.5 mmol microcrystalline KCl a total of 6000 mg of K in 2 EGJ, but split into 2 intakes daily) or PGJ for 28 days.

SUMMARY:
Rheumatoid arthritis is the paradigmatic immune-mediated inflammatory arthropathy. With respect to rheumatoid arthritis (RA), patients have been described as having inappropriately low spontaneous and stimulated cortisol secretion levels. Serum cortisol levels are decreased in RA patients who are taking prednisolone. Also, in patients RA, of longer duration, glucocorticoid receptor (GR) down-regulation has been reported without any change in cortisol levels. There is a reduced capacity for local reactivation of cortisone to cortisol in RA synovial cells. It is noteworthy that since synthetic glucocorticoids also use same reactivation shuttle (the cortisol-cortisone shuttle), the results also apply to therapeutic glucocorticoids.

Glucocorticoids are widely used to treat chronic inflammatory conditions including rheumatoid arthritis. Prednisolone has a greater effect than non-steroidal, anti-inflammatory drugs on joint tenderness and pain, whereas the difference in grip strength was not significant. There are no qualitative differences between the effects of endogenous cortisol and exogenously applied synthetic glucocorticoids, since all effects are transmitted via the same receptor. Cortisol, on the other hand, plays a major role in normal potassium homeostasis.

Recent studies have highlighted a role for diet, with suggestions that diets high in caffeine, low in antioxidants and high in red meat may contribute to an increased risk for the development of rheumatoid arthritis. Higher intakes of complex carbohydrates, dietary fiber, magnesium, folic acid, vitamin C and E, carotenoids and other phytochemicals have been shown to offer distinct advantages compared to diets containing meat and other foods of animal origin. The relation of a potassium deficiency to RA is much less well documented. The first person to definitively link potassium with arthritis was DeCoti Marsh. LaCelle, Morgan & Atwater found that the cells of 50 arthritic patients were 30 to 50% lower than healthy people.

Our current clinical trial (clinical trial no NCT00399282) shows that most of patients with RA do not have enough potassium intake. This condition may contribute to a subclinical lower serum cortisol, although there is possibility that cortisol serum levels might be unchanged due to a sufficient "cortisol homeostasis" and "potassium homeostasis".

DETAILED DESCRIPTION:
This study examines the hypothesis if patients with rheumatoid arthritis evaluate, or rate, symptom improvements after potassium supplementation (as KCl).

Participants will undergo the following tests and procedures:

Medical history and physical examination. Measurements of weight and height. Blood sample collections for clinical and research purposes. Quality of life questionnaires.

We therefore examined the hypothesis that examines effect of an orally administrated grape juice enriched (GJE) with 6000 mg potassium (as KCl) compared with that of a placebo grape juice (PGJ) on serum indices (cortisol, ACTH, aldosterone, creatinine, pH, Na, K), urinalysis (urea, uric acid, K, Na, creatinine, pH), GFR corrected by body surface area, ESR, CRP, RF, pain, quality of life, and disease activity in a case-controlled double-blind protocol in patients with RA with an established low dietary potassium intake to further investigate endogenous cortisol secretion and consequent possible relief.

Clinical (like Disease Activity, Pain) variables, along with the Quality of Life, and Biochemical Indices will be compared in two groups of patients after 28 days of oral GJE and PJE administration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of RA, as defined by fulfilling at least four of seven American College of Rheumatology (ACR) criteria
* Onset of arthritis after the age of 16 years
* Positive for rheumatoid factor (RF)
* Active RA, as defined by at least four swollen joints, at least four tender joints, and either an erythrocyte sedimentation rate (ESR) of greater than 30 mm/hr OR C-reactive protein level greater than 1.0 mg/dl (normal less than 0.4)
* Willing to follow the study protocol
* Willing to intake PGJ or EGJ
* On a salt-restricted diet

Exclusion Criteria:

* Abnormal kidney (including kidney stones in the 5 years prior to study entry or creatinine clearance less than 50 ml/min/1.73 m2 of body surface area) or liver disease
* Currently taking medications that might affect potassium
* Intra-articular injections within 4 weeks prior to study entry
* Current peptic ulcer disease
* History of alcohol or substance abuse
* Active infection, or chronic or persistent infection that might worsen with immunosuppressive treatment (e.g., HIV, hepatitis B virus, hepatitis C virus, tuberculosis [TB])
* Known coronary artery disease or significant cardiac arrhythmias or severe congestive heart failure (New York Heart Association [NYHA] classes III or IV)
* Definitive diagnosis of another autoimmune rheumatologic disease (e.g., systemic lupus erythematosus [SLE], scleroderma, primary Sjogren's syndrome, primary vasculitis)
* History of cancer. Participants with previous resected basal or squamous cell carcinoma, treated cervical dysplasia, or treated in situ Grade I cervical cancer within 5 years prior to study entry are not excluded.
* Any condition or treatment (including biologic therapies) that, in the opinion of the investigator, may place the participant at unacceptable risk during the study
* Pregnancy
* Vegetarian
* Use of estrogen replacement therapy
* Current use of diuretics, beta-blockers, anabolic drugs (steroids or other), angiotensin converting enzyme (ACE) inhibitors, or angiotensin receptor blockers (ARBs), etc, or any drug (s) other than drugs indicated for the purpose of RA therapy which is (are) known to effect serum potassium levels
* Hyperparathyroidism
* Untreated thyroid disease
* Significant immune disorder
* Adrenal insufficiency, primary aldosteronism, or Bartter's syndrome
* Diabetes mellitus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Patient's dietary and supplement potassium intake (combined technique: food frequency questionnaire, 24 hour food-recall, food record), serum potassium | within the 28 days (plus or minus 2 days)
Disease Activity Score (DAS28, 28-joint count) at d 0, 28 | within the first 28 days (plus or minus 2 days)
Patient's global assessment of disease activity (0 to 10 cm visual analog scale: 0, symptom free; 10, very severe) at d 0, 28 | within the first 28 days (plus or minus 2 days)
Patient's visual analogue scale (VAS) for pain at d 0, 28 | within the first 28 days (plus or minus 2 days)
Duration of morning stiffness (in minutes) at d 0, 28 | within the first 28 days (plus or minus 2 days)
Joint pain intensity, on a visual analogue scale (VAS) for pain (0 = no pain to 100mm =severe pain) at d 0, 28 | within the first 28 days (plus or minus 2 days)
Onset of fatigue (in minutes) after walking at d 0, 28 | within the first 28 days (plus or minus 2 days)
Ritchie's articular index for pain joints at d 0, 28 | within the first 28 days (plus or minus 2 days)
Right and left grip strength (in mmHg) measured with a sphygmomanometer cuff inflated to 20 mmHg at d 0, 28 | within the first 28 days (plus or minus 2 days)
Classification of functional status in RA according to revised criteria of the American College of Rheumatology at Patient's global assessment of disease activity (0 to 10 cm visual analog scale: 0, symptom free; 10, very severe) at d 0, 28 | within the first 28 days (plus or minus 2 days)

SECONDARY OUTCOMES:
Serum cortisol, NA, K, ACTH, aldosterone, creatinine, urea, uric acid, pH; urinalysis (urea, uric acid, Na, K, pH, creatinine), CRP, RF, and ESR at d 0, 28 | within the first 28 days (plus or minus 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Rastmanesh, Ph.D., Study Chair — National Nutrition and Food Sciences Technology Institute
Locations (2):
- Iran (2):
  - Division of Rheumatoloy, Sina Teaching Hospital, Tabriz Medical Sciences University, Tabriz, East Azerbaidjan
  - Sheikh-ol-Raees Ultra Specialized Clinic, Tabriz, East Azerbaidjan

REFERENCES:
- [Background] Weber CE. Copper response to rheumatoid arthritis. Med Hypotheses. 1984 Dec;15(4):333-48. doi: 10.1016/0306-9877(84)90150-6. PMID 6152006
- [Background] Weber CE. Corticosteroid regulation of electrolytes. J Theor Biol. 1983 Oct 7;104(3):443-9. doi: 10.1016/0022-5193(83)90116-9. PMID 6656267
- [Background] Weber CE. A proposal for an experiment of potassium on rheumatoid arthritis. Clin Exp Rheumatol. 1983 Apr-Jun;1(2):184-6. No abstract available. PMID 6398157
- [Result] Rastmanesh R, Abargouei AS, Shadman Z, Ebrahimi AA, Weber CE. A pilot study of potassium supplementation in the treatment of hypokalemic patients with rheumatoid arthritis: a randomized, double-blinded, placebo-controlled trial. J Pain. 2008 Aug;9(8):722-31. doi: 10.1016/j.jpain.2008.03.006. Epub 2008 May 12. PMID 18468955
- [Result] Rastmanesh R. Psoriasis and vegetarian diets: a role for cortisol and potassium? Med Hypotheses. 2009 Mar;72(3):368. doi: 10.1016/j.mehy.2008.09.031. Epub 2008 Nov 4. No abstract available. PMID 18986773
- See also: Related Info — http://www.clinicaltrials.gov/ct/show/NCT00399282?order=2